CLINICAL TRIAL: NCT03514095
Title: Cognitive Stimulation in the Elderly: Individual Intervention on Cognitive Frailty
Acronym: ECOG_CS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Escola Superior de Enfermagem de Coimbra (Other)
Collaborators: Grouping of Health Centers of Greater Porto I - Santo Tirso/Trofa (Other); Group of Health Centers of Greater Porto IV - Póvoa de Varzim/Vila do Conde (Other)
Responsible Party: Principal Investigator, Joao Apostolo, Ph.D, Coordinator Professo, Escola Superior de Enfermagem de Coimbra
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: ECOG_CS
Record Dates: First submitted 2018-04-20; First posted 2018-05-02 (Actual); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Neurocognitive Disorders; Dementia
MeSH Terms: conditions — Neurocognitive Disorders; Dementia

STUDY DESIGN:
Intervention Model Description: Participants will be assigned in two groups, a control group who will usual care by their caregivers and an experimental group who will receive the MD3 program.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The randomization process it will be done in https://www.random.org/ by an independent person.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): The control group shall participate in the usual home-based care provided by their carer.
- Individual Cognitive Stimulation Therapy (Experimental): The experimental group shall participate in the Making a Difference 3 program (Yates et al., 2015) is aimed at elderly people with mild or major neurocognitive disorder, where informal caregiver (family, friend or neighbour) assume a partnering role in an one-to-one approach. The program is composed by a range of stimulating activities (sessions), each with two levels of difficulty. The carers are introduced to a set of key principles that guides them during individual cognitive stimulation sessions, tailoring the interventions to the needs and reality of the elderly participants.
  Interventions: Other: Individual Cognitive Stimulation Therapy Program

INTERVENTIONS:
Other: Individual Cognitive Stimulation Therapy Program — This program unfolds in 3 weekly sessions of 30 minutes, for 12 weeks, thus completing a total of 36 sessions.
  Over the 3 months, the dyad will need to be monitored for orientation / monitoring of intervention by an element of the research team. This monitoring will be bi-weekly, in person or by phone - here according to the choice of the dyad). After each session the caregiver has a questionnaire to complete (intervention monitoring strategy), with the objective of evaluating the acceptability and applicability of the program.
  Arms: Individual Cognitive Stimulation Therapy

SUMMARY:
Cognitive Stimulation (CS) in the elderly, as a group intervention, shows benefits on the cognition and quality of life of people with neurocognitive disorder (NCD)(ie, dementia). The evidence of cognitive stimulation as an individualized intervention, conducted at home, by the caregiver is limited. The main objective of this trial is to evaluate the effectiveness of the Individual Cognitive Stimulation Therapy program - "Making a Difference 3 - individual Cognitive Stimulation Therapy (MD3), its acceptability and applicability by the dyad (people with NCD and their caregiver) in the Portuguese population. To achieve this purpose a pilot study will be conducted (randomized control trial), with two moments of evaluation - before the intervention of individual cognitive stimulation and after the intervention in both groups (Group 1 - group subject to intervention: individual cognitive stimulation program called "MD3"; Group 2 - group subject to usual care).The investigators intend to know the effect of the program on cognitive domains, quality of life and relationship between caregiver and care recipient. And, as well as understand the acceptability and applicability of the program by participants (dyad).

DETAILED DESCRIPTION:
Caring for people with mild and major neurocognitive disorder (NCD) is a major challenge for the current international health care systems. People with NCD lack care to meet their needs, which makes the development and implementation of specific interventions a priority. These should aim to increase the self-care potential of people with mild and major NCD, by promoting their autonomy and family support.

"Making a Difference 3 (MD3) - Individual Cognitive Stimulation Therapy: A manual for carers" is an example of an individual cognitive stimulation program. This program is useful for a large number of elderly people who, for various reasons, can not participate in group cognitive stimulation program. This individual cognitive stimulation can be developed in several settings, including in people's homes and with use of inexpensive resources, but very little knowledge has been produced in this area. Studies carried out in the family environment and involving the caregiver showed gains for the people, such as improvement in cognitive performance including memory, verbal fluency, problem solving capacity, less institutionalization; and for their caregivers, improvement in their overall well-being including decreased feelings of hostility.

However, the methodological fragility of these studies is emphasized in both the design, sample size and lack of uniformity in the type and time of the intervention. The individual cognitive stimulation that we intend to study by applying the MD3 program is considered a complex intervention because it followed in its construction the guidelines recommended by the Medical Research Council.

The efficacy study of this individual cognitive stimulation program, developed at the National Health Service (NHS) in England, and which we intend to replicate in part, was a 25-week randomized controlled trial of 273 dyads. In this study, there were no statistically significant differences between the experimental group and the control group in the outcomes evaluated as: cognition, self-report quality of life, psychological and behavioral symptomatology, and depressive symptomatology. Regarding the caregivers, the study revealed that there were no statistically significant differences in mental and physical health between groups, but the intervention group revealed a higher quality of life. However, some conditioning factors that may have compromised the final results of this study, namely the loss of participants and the low adherence to the program (22% of the participants did not complete any of the sessions and only 51% of the dyads completed more than 30 sessions). Dyads that completed more sessions showed improvement in the quality of the relationship, while the caregivers showed less depressive symptoms.

The investigators understand that, in the context of these results, more studies are needed to evaluate the effects of this program, but mainly it is necessary to find strategies that limit the low adherence and understand the applicability of the MD3 program.

In summary, there is no evidence base on the efficacy of individual cognitive stimulation in people with mild or major NCD in the home setting of the elderly, managed by the informal caregiver and supervised by health professionals (eg nurses). In addition, in Portugal, there are still no structured programs of cognitive stimulation with individual sessions for use in the home context. In this sense, the team of the present project proposes to produce national evidence on the efficacy of individual cognitive stimulation in people with mild and major NCD in the elderly domiciliary context, managed by the informal caregiver and supervised by health professionals. Simultaneously, to know the acceptability (by the adhesion - number of stimulation sessions performed - by the dyad) and the practicability of the program (evaluate to what extent the sessions are practical and practicable within the home context.

ELIGIBILITY:
Inclusion Criteria:

* Elderly person with 60 years of age or older;
* Diagnosis of mild or major neurocognitive disorder, performed by a physician specialized in neurology or psychiatry, or who is validated by the family physician in accordance with DSMIII/IV/5 or ICD-9/10 criteria;
* Presence of mild to moderate cognitive impairment according to the 6-Item Cognitive Decline Test (6CIT);
* Capable of communicating and understanding communication;
* Without a physical illness or significant disability (eg elderly people who are on dialysis or bedridden);
* Living in the community (in their home);
* Have an informal caregiver available and able to develop the individual cognitive stimulation program.

Exclusion Criteria:

* Elderly / informal caregiver with a history of severe psychiatric illness diagnosed before 60 years of age;
* Informal caregiver with cognitive impairment, even if mild (mild PNC according to DSM-5 criteria);
* Elderly people who do not live in their home.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-06-30 (Estimated); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the elderly participant's Cognition | Post-intervention assessment (week 13)
  Outcome Measure - Alzheimer's Disease Assessment Scale - Cognitive Subscale (Rosen et al., 1984).
Change from Baseline in the elderly participant's Quality of Life | Post-intervention assessment (week 13)
  Outcome Measure - Quality of Life in Alzheimer's Disease (Logsdon et al., 2002).
Change from Baseline in the caregiver's overall health | Post-intervention assessment (week 13)
  Outcome Measure - Short Form-12 Health Survey (Ware et al., 1996).

SECONDARY OUTCOMES:
Change from Baseline in the elderly participant's Neuropsychiatric Symptoms | Post-intervention assessment (week 13)
  Outcome Measure - The Neuropsychiatric Inventory Questionnaire(Cummings et al.,1994)
Change from Baseline in the elderly participant's Functional Capacity | Post-intervention assessment (week 13)
  Outcome Measure - Barthel Index of Activities of Daily Living (Mahoney & Barthel, 1965)
Change from Baseline in the elderly participant's Depressive Symptoms | Post-intervention assessment (week 13)
  Outcome Measure - Geriatric Depression Scale - 15 items (Sheikh & Yesavage,1986)
Change from Baseline in the dyad's (elderly participant and caregiver) Quality of the Relationship | Post-intervention assessment (week 13)
  Outcome Measure - Quality of the carer-patient relationship (Spruytte, 2002)

CONTACTS AND LOCATIONS:
Locations (1):
- Health Sciences Research Unit: Nursing, Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brooke P, Bullock R. Validation of a 6 item cognitive impairment test with a view to primary care usage. Int J Geriatr Psychiatry. 1999 Nov;14(11):936-40. PMID 10556864
- [Background] Yates, L.; Orrel M., Phoung, L.; Spector, O.; Woods, B.; Orgeta V. Making a Difference 3 - Individual Cognitive Stimulation Therapy: A manual for carers. London: The Journal of Dementia Care : Hawker Publications; 2015. 160 p.
- [Background] Spruytte N, Van Audenhove C, Lammertyn F, Storms G. The quality of the caregiving relationship in informal care for older adults with dementia and chronic psychiatric patients. Psychol Psychother. 2002 Sep;75(Pt 3):295-311. doi: 10.1348/147608302320365208. PMID 12396755
- [Background] Orgeta V, Leung P, Yates L, Kang S, Hoare Z, Henderson C, Whitaker C, Burns A, Knapp M, Leroi I, Moniz-Cook ED, Pearson S, Simpson S, Spector A, Roberts S, Russell IT, de Waal H, Woods RT, Orrell M. Individual cognitive stimulation therapy for dementia: a clinical effectiveness and cost-effectiveness pragmatic, multicentre, randomised controlled trial. Health Technol Assess. 2015 Aug;19(64):1-108. doi: 10.3310/hta19640. PMID 26292178
- [Background] Orrell M, Yates LA, Burns A, Russell I, Woods RT, Hoare Z, Moniz-Cook E, Henderson C, Knapp M, Spector A, Orgeta V. Individual Cognitive Stimulation Therapy for dementia (iCST): study protocol for a randomized controlled trial. Trials. 2012 Sep 22;13:172. doi: 10.1186/1745-6215-13-172. PMID 22998983
- [Background] Quayhagen, M. & Quayhagen, M. (2001). Testing of a cognitive stimulation intervention for dementia caregiving dyads. Neuropsychological Rehabilitation, 11(3), 319-332. http://doi.org/10.1080/09602010042000024
- [Background] Quayhagen MP, Quayhagen M, Corbeil RR, Hendrix RC, Jackson JE, Snyder L, Bower D. Coping with dementia: evaluation of four nonpharmacologic interventions. Int Psychogeriatr. 2000 Jun;12(2):249-65. doi: 10.1017/s1041610200006360. PMID 10937544
- [Background] Rosen WG, Mohs RC, Davis KL. A new rating scale for Alzheimer's disease. Am J Psychiatry. 1984 Nov;141(11):1356-64. doi: 10.1176/ajp.141.11.1356. PMID 6496779
- [Background] Logsdon RG, Gibbons LE, McCurry SM, Teri L. Assessing quality of life in older adults with cognitive impairment. Psychosom Med. 2002 May-Jun;64(3):510-9. doi: 10.1097/00006842-200205000-00016. PMID 12021425
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Cummings JL, Mega M, Gray K, Rosenberg-Thompson S, Carusi DA, Gornbein J. The Neuropsychiatric Inventory: comprehensive assessment of psychopathology in dementia. Neurology. 1994 Dec;44(12):2308-14. doi: 10.1212/wnl.44.12.2308. PMID 7991117
- [Background] MAHONEY FI, BARTHEL DW. FUNCTIONAL EVALUATION: THE BARTHEL INDEX. Md State Med J. 1965 Feb;14:61-5. No abstract available. PMID 14258950
- [Background] Sheikh, J. I., & Yesavage, J. A. (1986). Geriatric Depression Scale (GDS): Recent evidence and development of a shorter version. Clinical Gerontologist, 5, 165-173.
- [Derived] Silva R, Bobrowicz-Campos E, Santos-Costa P, Cruz AR, Apostolo J. A Home-Based Individual Cognitive Stimulation Program for Older Adults With Cognitive Impairment: A Randomized Controlled Trial. Front Psychol. 2021 Nov 22;12:741955. doi: 10.3389/fpsyg.2021.741955. eCollection 2021. PMID 34880809